## **Consent Cover Page**

Improving Health Insurance Literacy among Utah's Hispanic Community
HIEP Pilot—Hispanic Community Members

Approved by the University of Utah Institution Review Board on 03/10/2021 IRB\_00138483

## **Consent Cover Letter**

## Improving Health Insurance Literacy among Utah's Hispanic Community

HIEP Pilot – Hispanic Community Members

The purpose of this research study is to adapt and refine a health insurance education program to the Hispanic community in Utah. We are doing this study because Hispanics are more likely to be uninsured and often experience barriers accessing and using health insurance. This research study will help us refine educational materials specifically to help the Hispanic community understand and use their health insurance.

We would like to ask you to participate in a pilot test of our health insurance education program (HIEP). As part of this study, you will be asked to participate in the HIEP that was adapted to the Hispanic community, which involves going over the materials provided in the education program and completing short surveys regarding the education program to help us improve it moving forward. The HIEP pilot will be recorded for quality control purposes. A transcription service, will also have access to your information for transcribing your interview and all of this information will be kept secure and encrypted. There are minimal risks for participating in this study, but there is a slight chance for breach of confidentiality or discomfort while learning about health insurance. We will do everything possible to ensure the privacy and confidentiality of your responses.

We will also keep information you share in the survey or pilot from those not associated with the project. All electronic files will be kept on secured network drives and will be accessed via password-protected and encrypted computers by authorized members of the research team. Additionally, the information you provide in the survey or pilot will be kept in locked filing cabinets in a secure office, and will only be accessed by authorized members of the research team. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time

If you have any questions, complaints, or if you feel you have been harmed by this research please contact Dr. Anne Kirchhoff at the Huntsman Cancer Institute at 801-587-4084 or at <a href="mailto:anne.kirchhoff@hci.utah.edu">anne.kirchhoff@hci.utah.edu</a>.

Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

It should take approximately 2 hours to complete the HIEP pilot and about 20 minutes to complete the surveys. Participation in this study is voluntary. You can choose not to take part. You can choose not to finish the HIEP pilot and survey or omit any question you prefer not to answer without penalty.

By filling out this survey, you are giving your consent to participate.

We greatly appreciate your time and willingness to participate in this study. To thank you for your time and effort taking the pre and post surveys, we will give you two \$25 gift cards, one for each survey.

FOOTER FOR IRB USE ONLY Version: K0218



University of Utah Institutional Review Board Approved 3/10/2021

IRB\_00138483